CLINICAL TRIAL: NCT07400939
Title: Investigating The Neurophysiological Mechanisms Of Transcranial Direct Current Stimulation Combined With Action Observation Therapy On Hand Muscle Neuroplasticity in Chronic Stroke
Brief Title: Brain Stimulation Combined With Watching Hand Movements to Improve Hand Recovery in Chronic Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Malaysia Sabah (Other)
Responsible Party: Principal Investigator, Candace Goh Xiao Huey, Principal Investigator, Universiti Malaysia Sabah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMRR ID-24-00969-PKS
Record Dates: First submitted 2026-01-28; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Stroke; tDCS; Action Observation Therapy; Hand; Motor Evoked Potential; EMG; Neuroplasticity; Neurophysiological Assessment
Keywords: stroke rehabilitation; transcranial direct current stimulation; action observation therapy; neuroplasticity; neurophysiological
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active tDCS + AOT (Experimental): Participants will receive anodal transcranial direct current stimulation (tDCS) at 2 mA for 20 minutes combined with action observation therapy (AOT) for 10 sessions over 2 weeks at an outpatient clinic. During tDCS delivery, participants will observe first-person perspective videos of hand motor tasks and practice the observed movements. Following the clinic phase, participants will continue AOT practice at home for 30 minutes once daily for 8 weeks.
  Interventions: Other: tDCS; Other: Action Observation Therapy (AOT)
- sham tDCS + AOT (Placebo Comparator): Sham tDCS group - apply sham anodal tDCS with a 30s ramp-up and 30s ramp-down, switching the current to 0mA without the participant's awareness.
  Administer sham anodal tDCS for 20 minutes. Concurrently perform AOT for 30 minutes.
  Interventions: Other: Action Observation Therapy (AOT)
- tDCS only (Active Comparator): Administer active anodal tDCS for 20 minutes. Concurrently perform upper limb motor task actions with landscape video for 30 minutes.
  Interventions: Other: tDCS

INTERVENTIONS:
Other: tDCS — * Stimulation type: Anodal stimulation
  * Electrode size: 5x7cm
  * Stimulation target: C3/C4 primary motor cortex (M1) based on the 10-20 international electroencephalography system
  * Stimulation intensity: 2 mA
  * Stimulation current density: 0.029-0.057 mA/cm2
  Use tDCS with two saline-soaked surface sponge electrodes (5x7cm) applied to the scalp, secured with a headband. Stimulation intensity is set to 2mA, with 30s ramping up at the start and 30s ramping down at the end of stimulation.
  Arms: Active tDCS + AOT; tDCS only
Other: Action Observation Therapy (AOT) — Participants watch selected videos based on muscle grading of triceps, which include functional movement patterns and daily activity tasks of the upper limb. These videos are presented through a computer or mobile screen positioned at an appropriate distance from the participant to allow ample space for performing the required movements.
  Arms: Active tDCS + AOT; sham tDCS + AOT

SUMMARY:
This study investigates the neurophysiological and electrophysiological mechanisms underlying the combined use of transcranial direct current stimulation (tDCS) and action observation therapy (AOT) for hand motor recovery in individuals with stroke. Background: While both tDCS and AOT have shown promise individually for stroke rehabilitation, the neural mechanisms of their combined effects remain unclear. Understanding these mechanisms could optimise rehabilitation protocols and improve functional outcomes. Intervention: Participants will receive 10 sessions of anodal tDCS over the ipsilesional motor cortex combined with AOT over two weeks in a clinical setting, followed by 8 weeks of home-based AOT practice. Control groups will receive tDCS alone or AOT alone. Neurophysiological changes will be assessed using motor evoked potentials (MEPs) to evaluate corticospinal excitability. Clinical hand function will be assessed using standardised outcome measures. Measurements: Assessments will be conducted at baseline, during intervention (week 2), and after the home practice phase (week 10) to evaluate neuroplastic changes. Significance: This study will provide mechanistic insights into how neuromodulation and observational learning interact to promote motor recovery, informing evidence-based rehabilitation strategies for stroke survivors in Malaysia and globally. Study Design: Randomised controlled trial with three parallel arms, recruiting 60 participants with chronic stroke from Sabah, Malaysia.

DETAILED DESCRIPTION:
The participation duration for each participant is 10 weeks, including the assessment period.

Group 1 tDCS + AOT (intervention): tDCS will be administered at the outpatient clinic for 20 minutes per session, for a total of 10 sessions over two consecutive weeks. During the tDCS sessions, each participant will engage in AOT for 30 minutes under the supervision of a therapist. Subsequently, each participant will continue performing AOT at home for 30 minutes per session, once a day, five days per week, for 8 consecutive weeks.

Group 2 tDCS alone (control): tDCS will be administered at the outpatient clinic for 20 minutes per session, for a total of 10 sessions over two consecutive weeks. During the tDCS sessions, each participant will watch a landscape video for 30 minutes. Subsequently, each patient will continue watching the landscape video at home for 30 minutes per session, once a day, five days per week, for 8 consecutive weeks.

Group 3 AOT alone (control): placebo tDCS will be administered at the outpatient clinic for 20 minutes per session, for a total of 10 sessions over 2 consecutive weeks. During the placebo tDCS sessions, each participant will engage in AOT for 30 minutes under the supervision of a therapist. Following the clinic sessions, each patient will continue performing AOT at home for 30 minutes per session, once a day, five days per week, for 8 consecutive weeks.

The principal investigator will visit each research site throughout the duration of the study. All participants will attend the outpatient rehabilitation setting five times a week for 30 minutes per session, for 2 consecutive weeks, and continue intervention at home for five days a week for 8 consecutive weeks. The total intervention duration consists of 10 consecutive weeks. For each session in the hospital, there will be a physiotherapist to monitor participants' compliance with the interventions and to ensure that the training is conducted as per protocol. Level of participation would be measured by Rating of Perceived Exertion Scale of 3-5 (light activity to somewhat hard). If the subject attended the session but refuse to participate in the intervention, the subject would be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 59 years
* Single episode of unilateral stroke and weakness in hand muscles 6 to 24 months post-stroke
* No excessive spasticity of the upper limb, defined as grade two or less on Modified Ashworth Scale

Exclusion Criteria:

* Patients diagnosed with posterior circulation infarction
* Unable to follow commands due to poor cognitive function
* Unilateral neglect
* Homonymous hemianopia
* Other existing neurological disorders that lead to poor hand function
* Grade four or five hand muscle strength.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-01-20 (Estimated); Study Completion 2028-01-20 (Estimated)

PRIMARY OUTCOMES:
Motor Evoked Potentials (MEPs) | From enrolment to the end of treatment at 10 weeks
  Peak-to-peak amplitude of motor evoked potentials (MEPs) elicited by single-pulse transcranial magnetic stimulation (TMS) and recorded via surface electromyography (EMG) from hand muscles of the paretic upper limb.
  Assessment Method:
  * TMS delivers single pulses over ipsilesional primary motor cortex (M1 hand area)
  * Surface EMG electrodes record responses from first dorsal interosseous (FDI), abductor pollicis brevis (APB), and extensor carpi radialis (ECR) muscles
  * Motor hotspot identified (optimal scalp location producing largest MEPs)
  * Resting motor threshold determined
  * 15-20 MEPs recorded at 120% of resting motor threshold
  * Inter-stimulus interval: 5-7 seconds
  * MEP amplitude measured as peak-to-peak voltage in millivolts (mV)

CONTACTS AND LOCATIONS:
Overall Officials: Fatimah Ahmedy, Principal Investigator — Universit Malaysia Sabah
Locations (3):
- Malaysia (3):
  - Beaufort Hospital, Beaufort, Sabah
  - Hospital Universiti Malaysia Sabah (HUMS), Kota Kinabalu, Sabah
  - Queen Elizabeth Hospital, Kota Kinabalu, Sabah